CLINICAL TRIAL: NCT01224470
Title: The Effects of Intravenous Dexmedetomidine on Spinal Anesthesia Using Low Dose Diluted Bupivacaine for Transurethral Resection of Prostate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Hae Keum Kil / Professor, Anesthesiology and Pain Medicine, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 4-2010-0405
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Transurethral Prostatectomy
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bupivacaine (Active Comparator): 0.5% bupivacaine 1.2 mL + normal saline 0.8 mL = total 2 mL
  Interventions: Drug: Dexmedetomidine
- saline (Placebo Comparator)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexamedetomidine intravenous injection (1 ㎍/kg )
  Other Names: brand name : PRECEDEX; (generic name : Dexmedetomidine)

SUMMARY:
Dexmedetomidine is a new selective and potent alpha-2 agonist. It has centrally acting anesthetic properties. It has been known that intrathecal addition of alpha-2 adrenergic agents result in prolongation of the duration of the sensory and motor blockade induced by hyperbaric bupivacaine. But the effects of intravenous dexmedetomidine on the spinal block was not evaluated. The aim of study is to assess the effect of intravenous dexmedetomidine on the low-dose spinal anesthesia for the transurethral surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I or II
* Elective transurethral prostatectomy
* aged > 20

Exclusion Criteria:

* Coagulation deficiency
* infection on the back
* Congestive heart failure or arrythmia
* Chronic alcoholic disease
* Antidepressants therapy

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-11; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Hong JY, Kim WO, Yoon Y, Choi Y, Kim SH, Kil HK. Effects of intravenous dexmedetomidine on low-dose bupivacaine spinal anaesthesia in elderly patients. Acta Anaesthesiol Scand. 2012 Mar;56(3):382-7. doi: 10.1111/j.1399-6576.2011.02614.x. Epub 2012 Jan 4. PMID 22220945